CLINICAL TRIAL: NCT04668820
Title: Reliability and Acceptability of Real-time Virtual Video Pediatric Gait, Arms, Legs and Spine (V-pGALS) Assessment for Musculoskeletal Assessment of Children for Telemedicine Visits
Brief Title: Reliability and Acceptability of Real-time Virtual Video Pediatric Gait, Arms, Legs and Spine (V-pGALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09.2020.1
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-12

CONDITIONS: Musculoskeletal Abnormality; Pediatric
Keywords: telemedicine; pandemic; video Pediatric Gait, Arms, Legs and Spine (V-pGALS); pediatric examination; musculoskeletal examination; reliability; acceptability
MeSH Terms: conditions — Musculoskeletal Abnormalities; Rhabdomyosarcoma, Alveolar

STUDY DESIGN:
Intervention Model Description: Children between the ages of 7-18 who admit pediatric rehabilitation outpatient clinic
Masking Description: Two phsyiatrist who will perform virtual video Pediatric Gait, Arms, Legs and Spine (V-pGALS) and the physiatrist who will perform face to face examination will be blinded to each other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children who admit to Pediatric Rehabilitation outpatient clinic (Experimental): Children who admit to Pediatric Rehabilitation outpatient clinic of the Department of Physical Medicine and Rehabilitation will be evaluated by face to face and virtually by using zoom application via video Pediatric Gait, Arms, Legs and Spine (V-pGALS)
  Interventions: Diagnostic Test: video Pediatric Gait, Arms, Legs and Spine (V-pGALS)

INTERVENTIONS:
Diagnostic Test: video Pediatric Gait, Arms, Legs and Spine (V-pGALS) — The Video-pGALS includes maneuvers from pediatric regional examination of the musculoskeletal system (pREMS) and derived from the pediatric gait arms legs spine examination assessment which is a validated simple basic musculoskeletal (MSK) examination for children. V-pGALS offers a structured approach to a cursory overview MSK exam with a focus on range of movement and symmetry. Utilizing the parent or caregiver to feel the joint in question for obvious warmth/ swelling or to palpate for point of maximal tenderness can add important information.

SUMMARY:
The use of telemedicine in musculoskeletal assessment has been historically low. The current COVID 19 global pandemic has forced a paradigm shift with many centers rapidly adopting virtual visits to conduct care resulting in rapid expansion of use of telemedicine amongst practices. Mayoclinic has published The Telemedicine Musculoskeletal Examination for adults. Paediatric Musculoskeletal Matters (PMM) has put video Pediatric Gait, Arms, Legs and Spine (V-pGALS) assessment sheet on their website. However, there is a lack of the acceptability and reliability of these tools. The aim of this study is to investigate acceptability and reliability of real-time virtual video Pediatric Gait, Arms, Legs and Spine (V-pGALS) assessment for musculoskeletal assessment of children for telemedicine visits.

DETAILED DESCRIPTION:
The use of telemedicine in musculoskeletal assessment has been historically low. The current COVID 19 global pandemic has forced a paradigm shift with many centers rapidly adopting virtual visits to conduct care resulting in rapid expansion of the use of telemedicine amongst practices. Mayoclinic has published The Telemedicine Musculoskeletal Examination for adults. 'Paediatric Musculoskeletal Matters' (PMM- www.pmmonline.org, is a free, evidence-based, and peer-reviewed open e-resource for pediatric musculoskeletal (MSK) medicine targeting non-MSK specialists. They have also published video Pediatric Gait, Arms, Legs and Spine (V-pGALS), an assessment sheet for telemedicine visits on their webpage. However, there is a lack of the acceptability and reliability of these tools. The aim of this study is to investigate acceptability and reliability of real-time virtual video Pediatric Gait, Arms, Legs and Spine (V-pGALS) assessment for musculoskeletal assessment of children for telemedicine visits. For this purpose, children at between the ages of 7-18 who admitted the Pediatric Rehabilitation outpatient clinic of Department of Physical Medicine and Rehabilitation of Marmara University School of Medicine will be recruited to the study. They will be evaluated via V-pGALS face to face on the day of admission and the physiatrist will record the diagnosis if there is. Within 24 hours the child will be reevaluated via V-pGALS by using Zoom application virtually. The acceptability of V-pGALS examination to the child and parents in terms of the duration and additional discomfort caused was evaluated using visual analog scale with smiley faces (0-10, 0 for full acceptability).

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 7-18 who admitted the Pediatric Rehabilitation outpatient clinic of Department of Physical Medicine and Rehabilitation

Exclusion Criteria:

* Non-ambulatory children
* Children with poor cooperation
* Being severe ill and unable to tolerate examination
* Children and parents who do not give oral and written permission for study enrollment

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Face to face examination of video Pediatric Gait, Arms, Legs and Spine (V-pGALS) | Day 0
  Face to face examination
real-time virtual video Pediatric Gait, Arms, Legs and Spine (V-pGALS) | Day 1
  Video real-time examination via zoom application

SECONDARY OUTCOMES:
Acceptability of V-pGALS examination to the child in terms of the duration | Day 1
  visual analog scale with smiley faces (0-10, 0 for full acceptability)
Acceptability of V-pGALS examination to the child in terms of the additional discomfort caused | Day 1
  visual analog scale with smiley faces (0-10, 0 for full acceptability).
  visual analog scale with smiley faces (0-10, 0 for full acceptability).
  visual analog scale with smiley faces (0-10, 0 for full acceptability). visual analog scale with smiley faces (0-10, 0 for full acceptability).
  visual analog scale with smiley faces (0-10, 0 for full acceptability)
Acceptability of V-pGALS examination to the parent who will be present during examination in terms of the duration | Day 1
  visual analog scale with smiley faces (0-10, 0 for full acceptability)
Acceptability of V-pGALS examination to the parent who will be present during examination in terms of the additional discomfort caused | Day 1
  visual analog scale with smiley faces (0-10, 0 for full acceptability)

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag-Saygı, Prof, Study Chair — Marmara University School of Medicine Department of Physical Medicine and Rehabilitation; Esra Giray, assoc. prof, Principal Investigator — Koc University School of Medicine Department of Physical Medicine and Rehabilitation; Özden Ozyemisci Taskiran, Prof, Principal Investigator — Koc University School of Medicine Department of Physical Medicine and Rehabilitation; Ozge Kenis-Coskun, assoc. prof, Principal Investigator — Marmara University School of Medicine Department of Physical Medicine and Rehabilitation
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study will be available on request from the corresponding author (EG). The data will not be publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Batu ED, Kenis Coskun O, Sonmez HE, Karali D, Arslanoglu Aydin E, Bilginer Y, Karadag Saygi E, Ozen S. Acceptability and Practicality of the Turkish Translation of Pediatric Gait Arm Legs and Spine in Turkish Children. J Clin Rheumatol. 2017 Dec;23(8):421-424. doi: 10.1097/RHU.0000000000000586. PMID 28926470
- [Result] Pelaez F, de Haro C. Translational inhibition by eIF-2-phospholipid complex in mammalian cell-free systems. FEBS Lett. 1989 Jul 3;250(2):523-8. doi: 10.1016/0014-5793(89)80789-6. PMID 2753146
- [Result] Shenoi S, Hayward K, Curran ML, Kessler E, Mehta JJ, Riebschleger MP, Foster HE. Telemedicine in pediatric rheumatology: this is the time for the community to embrace a new way of clinical practice. Pediatr Rheumatol Online J. 2020 Oct 31;18(1):85. doi: 10.1186/s12969-020-00476-z. PMID 33129319
- [Derived] Giray E, Kenis-Coskun O, Karadag-Saygi E, Ozyemisci-Taskiran O. Interrater Reliability, Acceptability, and Practicality of Real-Time Video Pediatric Gait, Arms, Legs, and Spine for Musculoskeletal Assessment of Children During Telemedicine Visits. J Clin Rheumatol. 2022 Aug 1;28(5):235-239. doi: 10.1097/RHU.0000000000001840. Epub 2022 Mar 22. PMID 35319535